CLINICAL TRIAL: NCT04953286
Title: Tear Fluid and Ocular Surface Metabolomics and Lipidomics in Lateral Amyotrophic Sclerosis: a Prospective Comparative Study
Brief Title: Ocular Surface Metabolo-lipidomics in Lateral Amyotrophic Sclerosis
Acronym: LARMOMIQUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DR210051
Record Dates: First submitted 2021-05-17; First posted 2021-07-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2023-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Biomarkers; Ocular Surface; Tear
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Lacerations | interventions — Interferometry; Slit Lamp

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Other): The procedure, specific to the study, consists in taking samples of tears and cells at inclusion, 3 months after inclusion and 6 months after inclusion on patients with Amyotrophic Lateral Sclerosis
  Interventions: Other: Measure of visual acuity; Other: Interferometry; Other: Samples of basal tears; Other: Central corneal sensitivity; Other: Slit lamp examination and undilated fundus; Other: Conjunctival impression; Other: Evaluation of the corneal innervation
- Control group (Other): The procedure, specific to the study, consists in taking samples of tears and cells at inclusion, 3 months after inclusion and 6 months after inclusion on patients without neurological disease
  Interventions: Other: Measure of visual acuity; Other: Interferometry; Other: Samples of basal tears; Other: Central corneal sensitivity; Other: Slit lamp examination and undilated fundus; Other: Conjunctival impression; Other: Evaluation of the corneal innervation

INTERVENTIONS:
Other: Measure of visual acuity — ETDRS and Parinaud scale
Other: Interferometry — Non-contact exam measuring N.I.B.U.T (Non-invasive break-up time), quantitative and qualitative evaluation of the meibomian glands and quantitative evaluation of the tear meniscus
Other: Samples of basal tears — Collection of basal tears without instillation of anesthetic with a Schirmer strip for 5 minutes and by microcapillary
Other: Central corneal sensitivity — Central corneal sensitivity using a Cochet-Bonnet esthesiometer (Luneau©)
Other: Slit lamp examination and undilated fundus — Slit lamp examination and undilated fundus
Other: Conjunctival impression — Conjunctival impression with anesthetic instillation
Other: Evaluation of the corneal innervation — Contact corneal confocal microscopy

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is the most common neurodegenerative disease affecting the motor neuron. Currently, there is no diagnostic test and no examination that can predict the evolution of this pathology. The search for diagnostic and prognostic biomarkers is therefore essential for a better understanding of the pathophysiology of ALS, which remains poorly understood, and also for better clinical management. The ocular surface, made up of liquid elements, tears, and cells, is an accessible anatomical-physiological entity that has demonstrated its usefulness in the identification of biomarkers in neurodegenerative diseases such as Parkinson's or Alzheimer's. To date, no study has explored the ocular surface as a biomarker in ALS

ELIGIBILITY:
Case group selection criteria :

Inclusion Criteria:

* Patient with clinically defined or probable primary ALS according to Airlie House criteria(1)
* Familial or sporadic form
* ≥18 years of age
* Patient affiliated with a social security plan
* Informed consent signed by the patient

Exclusion Criteria:

* Motor neuron disease mimicking ALS
* Pregnant or breastfeeding woman
* Treatment that may have a neuroprotective effect
* Any eye drops or treatments that may interfere with tear production
* Lens wearer
* Eye surgery ≤3 months
* Any ocular pathology other than ametropia, oculomotor disorder, amblyopia
* Any general pathology other than ALS with ocular repercussions
* Protective measure of guardianship or curators

Control group selection criteria:

Inclusion Criteria:

* No diagnosed neurological pathology
* ≥18 years of age
* Patient affiliated with a social security plan
* Informed consent signed by the participant

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Treatment likely to have a neuroprotective effect
* Any eye drops or treatments that may interfere with tear production
* Lens wearer
* Eye surgery ≤3 months
* Any ocular pathology except ametropia, oculomotor disorder, amblyopia
* Any general pathology with ocular repercussions
* Protective measure of guardianship or curator

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Metabolome profile in tears for the diagnosis and prognosis of ALS. | Baseline
  Once the composition in metabolites (i.e. tear metabolome) is determined, statistical univariate and multivariate analyses will aim to determine if the tear metabolome can cluster ALS patients and controls and therefore can be used as a diagnosis biomarker
Metabolome profile in intra-cellular contents for the diagnosis and prognosis of ALS. | Baseline
  Once the composition in metabolites in conjunctival cells is determined, statistical univariate and multivariate analyses will aim to determine if the tear metabome can cluster ALS patients and controls and therefore can be used as a diagnosis biomarker.
Lipidome profile in tears for the diagnosis and prognosis of ALS. | Baseline
  Once the composition in lipids (i.e. tear lipidome) is determined, statistical univariate and multivariate analyses will aim to determine if the tear lipidome can cluster ALS patients and controls and therefore can be used as a diagnosis biomarker
Lipidome profile in intra-cellular contents for the diagnosis and prognosis of ALS. | Baseline
  Once the composition in lipids in conjunctival cells is determined, statistical univariate and multivariate analyses will aim to determine if the tear lipidome can cluster ALS patients and controls and therefore can be used as a diagnosis biomarker.

SECONDARY OUTCOMES:
Evolution of the ocular surface metabolites during ALS progression using ultra-high performance liquid chromatography coupled with mass spectrometry | Baseline
  By carrying out a longitudinal analysis in ALS cases, the modification in tear and cells metabo-lipidome will be assessed at three time-points (at diagnosis, at month 3 and 6) and will correlated with bioclinical criteria of ALS progression (i.e. % of weight loss, % of slope of progression of the ALS-FRS-r score and % of decrease in forced vital capacity). This analysis will aim to search for analytes that can predict ALS progression (i.e. prognosis biomarker).
Evolution of the ocular surface lipids during ALS progression using ultra-high performance liquid chromatography coupled with mass spectrometry | Baseline
  By carrying out a longitudinal analysis in ALS cases, the modification in tear and cells metabo-lipidome will be assessed at three time-points (at diagnosis, at month 3 and 6) and will correlated with bioclinical criteria of ALS progression (i.e. % of weight loss, % of slope of progression of the ALS-FRS-r score and % of decrease in forced vital capacity). This analysis will aim to search for analytes that can predict ALS progression (i.e. prognosis biomarker).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Ophthalmology Department, University Hospital of Tours, France, Tours
  - Neurology Department, University Hospital of Tours, France, Tours
  - Centre d'Investigation Clinique_CIC 1415, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khanna RK, Catanese S, Mortemousque G, Dupuy C, Lefevre A, Emond P, Beltran S, Gissot V, Pisella PJ, Blasco H, Corcia P. Metabolomics of basal tears in amyotrophic lateral sclerosis: A cross-sectional study. Ocul Surf. 2024 Oct;34:363-369. doi: 10.1016/j.jtos.2024.09.005. Epub 2024 Sep 28. PMID 39349171